CLINICAL TRIAL: NCT06390683
Title: Biodiversity Interventions for Well-Being - Research in Assisted Living Centers
Brief Title: Biodiversity Interventions for Assisted Living Centers
Acronym: BIWE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Resources Institute Finland (Other Government)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS/11940/2022
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Nature, Human; Microbial Colonization; Well-Being, Psychological; Immune System and Related Disorders; Autism Spectrum Disorder; Visual Impairment
Keywords: Biodiversity; Well-being; Planetary health; Commensal microbiome; Immune system
MeSH Terms: conditions — Communicable Diseases; Psychological Well-Being; Autism Spectrum Disorder; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rewilding (Experimental): Yards of the housing units are rewilded with vegetation, deadwood and plant residuals.
  Interventions: Other: Rewilding

INTERVENTIONS:
Other: Rewilding — Yards of the assisted living centers will be modified with berry bushes, fruit trees, perennial yard plants, meadow flowers, cultivation boxes, organic mulch materials, decaying deadwood, leaf compost and organic plant growing media with high microbial diversity.

SUMMARY:
Biodiversity is essential for nature and human well-being. Land use has reduced biodiversity in cities, which weakens the functionality of the urban ecosystems and the well-being of citizens. This may also increase the risk of immune-mediated disorders among urban dwellers.

In Biodiversity interventions for assisted living centers (BIWE 2), microbial biodiversity interventions are performed to increase biodiversity in urban housing units for people with autism spectrum disorder, disabled people and elderly. Results from the intervention trials are combined with publicly available land cover and ecological data. These are analyzed from the viewpoint of shifts in ecosystems and human well-being and immune regulation, ecological quality, and urban planning.

The investigators set up an intervention study in which yards of the housing units are rewilded with diverse vegetation and decaying deadwood and plant residuals. The investigators aim to evaluate the effect of rewilding, and yard management practices on commensal microbiome, cortisol levels and well-being and salivary cytokine levels, and gene pathways.

DETAILED DESCRIPTION:
Our specific aims are:

To assess if rewilding diversifies health-associated skin microbiota and is associated with salivary cytokine levels, gene pathways, cortisol levels and commensal microbiota.

Assess whether there are patterns in the microbiome associated with the salivary cytokine levels and hair cortisol levels.

Assess whether rewilding affects health and psychological measures. The investigators will recruit approximately 36 study subjects living in assisted housing units in urban areas and aged between 18-82.

ELIGIBILITY:
Inclusion Criteria:

* Person lives in assisted living center

Exclusion Criteria:

* Immunosuppressive medications
* Immune deficiencies
* a disease affecting immune response (colitis ulcerosa, rheumatoid arthritis, Crohn's disease, diabetes)
* cancer diagnosis within the last year or on-going cancer treatment

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Skin Gammaproteobacteria | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Change in skin gammaproteobacterial diversity

SECONDARY OUTCOMES:
Salivary cytokines | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Interleukin-6 and -10 measured from saliva
Skin bacteria | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Changes in skin bacteria are analyzed with Illumina 16s rRNA sequencing.
Saliva microbiota | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Changes in saliva microbiota are analyzed with shotgun sequencing.
Saliva gene pathways | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Changes in salivary gene pathways are analyzed with shotgun sequencing.
Cortisol levels | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Cortisol levels measured from hair samples
Perceived Stress Scale | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Decrease in perceived stress scale score during the study period that indicates lower perceived stress levels. Minimum 0, maximum 40.
Warwick-Edinburgh Mental Wellbeing Scale | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Increase in Warwick-Edinburhg Mental Wellbeing scale score during the study period that indicates better mental well-being. Minimum 14, maximum 70.
Depression Scale | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Decrease in depression scale score during the study period that indicates lower levels of depression symptoms. Minimum 0, maximum 70.
Nature Relatedness Scale | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Increase in Nature Relatedness scale during the study period that indicates stronger sense of connectedness to nature. Minimum 6, maximum 30.
Changes in nature contacts | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Increase in time that study subjects are in contact with nature during the study period.
Infectious diseases | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  Infectious diseases are recorded with questionnaires.

OTHER OUTCOMES:
Associations between environmental factors and primary and secondary outcomes | Baseline, 3 month, 1 year, 2 year, 3 year, 4 year, 5 year
  associations between environmental factors (vegetation, deadwood, and polypore richness, land cover categories and other yard characteristics), yard management practices, activities at the yard, salivary cytokine and hair cortisol levels, prevalence of infectious diseases, psychological parameters, and microbial measurements (diversity, and taxonomic and functional features).

CONTACTS AND LOCATIONS:
Overall Officials: Aki Sinkkonen, Principal Investigator — Natural Resources Institute Finland
Locations (1):
- Natural Resources Institute Finland, Helsinki, Uusimaa, Finland